CLINICAL TRIAL: NCT06749236
Title: A Single-center, Randomized, Open-label, Two-period, Crossover Clinical Study to Evaluate the Bioavailability of Two Specifications of Oral Deuterium Deuremidevir for Hydrobromide Suspension in Chinese Healthy Adult Participants
Brief Title: A Study to Evaluate the Bioavailability of Two Specifications of Oral Deuremidevir Hydrobromide for Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VV116-RSV-03
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test formulation(T) then reference formulation (R) of deuteriumremidvir hydrobromide for suspension (Experimental): On day 1 of the 1st period, participants will receive a single dose of the test formulation(T) (one bag of 200 mg deuteriumremidvir hydrobromide for suspension), and on day 1 of the 2nd period, participants will receive a single dose of the reference formulation(R) ( two bags of 100 mg deuteriumremidvir hydrobromide for suspension).The two periods are separated by a washout of 3 days.
  Interventions: Drug: test formulation(T) 200 mg deuteriumremidvir hydrobromide for suspension; Drug: reference formulation(R) 100 mg deuteriumremidvir hydrobromide for suspension
- reference formulation (R) then test formulation(T) deuteriumremidvir hydrobromide for suspension (Experimental): On day 1 of the 1st period, participants will receive a single dose of the reference formulation(R) ( two bags of 100 mg deuteriumremidvir hydrobromide for suspension), and on day 1 of the 2nd period, participants will receive a single dose of the test formulation(T) (one bag of 200 mg deuteriumremidvir hydrobromide for suspension).The two periods are separated by a washout of 3 days.
  Interventions: Drug: test formulation(T) 200 mg deuteriumremidvir hydrobromide for suspension; Drug: reference formulation(R) 100 mg deuteriumremidvir hydrobromide for suspension

INTERVENTIONS:
Drug: test formulation(T) 200 mg deuteriumremidvir hydrobromide for suspension — Participants will receive a single dose of the test formulation(T) (one bag of 200 mg deuteriumremidvir hydrobromide for suspension).
Drug: reference formulation(R) 100 mg deuteriumremidvir hydrobromide for suspension — Participants will receive a single dose of the reference formulation(R) ( two bags of 100 mg deuteriumremidvir hydrobromide for suspension).

SUMMARY:
The goal of this clinical study is to evaluate the bioavailability of two specifications of oral Deuteriumremidvir Hydrobromide for suspension in Chinese healthy adult participants. A total of 18 participants are planned to be enrolled and randomized into T-R or R-T sequence, 9 in each sequence with a single fasting administration in each period.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, two-period, crossover clinical study to evaluate the bioavailability of two specifications of oral deuteriumremidvir hydrobromide for suspension. With a washout period of 3 days, the dose is 200 mg in each sequence. The specification of the test formulation(T) is 200 mg and that for the reference formulation (R) is 100 mg. A total of 18 participants are planned to be enrolled and randomized into T-R or R-T sequence, 9 in each sequence with a single fasting administration in each period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old, males or females;
2. Male weight no less than 50 kg, female weight no less than 45 kg, body mass Index of 19 to 26 kg/m^2;
3. Vital signs examination, physical examination, laboratory examination and electrocardiogram examination results were normal or considered abnormal without clinical significance by the investigator;
4. Subjects who are willing to take proper contraceptive during the study and within 3 months after the the last administration;
5. Subjects who are able to understand and follow the study protocol and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. Participants with hypersensitivity to deuremidevir hydrobromide for suspension or any of the excipients;
2. Participants with allergic constitution (such as asthma, urticaria, eczematous dermatitis and other allergic diseases), or have a history of drug or food allergy;
3. Participants with central nervous system, cardiovascular system, gastrointestinal, respiratory system, urinary, hematologic, or metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
4. Participants who undergone surgery within 3 months before screening, or are planning to operate during the trial, or those who have undergone surgery that will affect the absorption, distribution, metabolism or excretion of drugs;
5. Participants who have received blood transfusion or used blood products within 3 months before screening or who have lost more than ≥400 mL of blood due to other reasons (except female physiological blood loss);
6. Participants who have participated in clinical trials of other drugs and received drugs within 90 days before screening;
7. Participants who have received vaccination within the first 1 month before screening, or planned to receive any vaccine during the trial or within 1 week after the end of the study；
8. Participants who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products orally within 2 weeks before screening;
9. Participants who have eaten grapefruits, pomelos, oranges, etc. within 7 days before screening, or do not agree to stop consuming the above fruits and drinks during the period;
10. Participants with a history of drug abuse within 1 year before screening or positive urine drug screening within 1 year before screening results (morphine, THC, methamphetamine, dimethylene diphetamine, ketamine, and cocaine);
11. Participants who drinking more than 14 standard units per week within one year before screening,(one standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of strong liquor with 40% alcohol content or 150 mL of wine), or being positive in the alcohol breath tests;
12. Participants who smoked more than 5 cigarettes a day within one year before screening;
13. Participants who can't quit smoking or drinking during the trial period;
14. Participants who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum antibody or human immunodeficiency virus antibody (Anti-HIV);
15. Abnormal chest X-ray results with clinical significance;
16. Abnormal ECG at screening or baseline, including QTcF (after heart rate correction) is >450 ms for males and > 470 ms for females in single examinations, and/or other abnormalities with clinical significance;
17. Participants who cannot tolerate blood collection with intravenous indwelling needles or blood fainting with dizzy needle;
18. Participants who cannot comply with a uniform diet (such as special dietary requirements, intolerance of standard meals, etc.), or be with lactose intolerance, or dysphagia;
19. Pregnant or lactating women or male participants whose spouse has a child care plan within 3 months;
20. The investigator believes that there are other unsuitable factors for this volunteer to participate this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Cmax | 48 hours after administration
  maximum observed plasma concentration
AUC0-t | 48 hours after administration
  area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | 48 hours after administration]
  area under the plasma concentration-time curve from time zero to infinity

SECONDARY OUTCOMES:
AUC0-24h | 24 hours after administration
  area under the plasma concentration-time curve from 0 to 24 hours
Tmax | 48 hours after administration
  time at which Cmax occurs
Tlag | 48 hours after administration
  time lag
t1/2 | 48 hours after administration
  half life of elimination
CLz/F | 48 hours after administration
  apparent clearance
Vz/F | 48 hours after administration
  apparent volume of distribution during the terminal phase
λz | 48 hours after administration
  first-order rate constant associated with the terminal (log-linear) portion of the curve
MRT | 48 hours after administration
  mean residence time
AE & SAE | from day1 to day6 after administration
  Adverse event & serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Xuzhou, Jiangsu, China